CLINICAL TRIAL: NCT03751930
Title: Intestinal Microbiota, Tryptophan and Autism
Acronym: MTA
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: DR180136; 2018-A01086-49 (Other: IdRCB)
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Tryptophan metabolism; Gut microbiota
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Sampling Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urinary and faecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Autism Spectre Disorders: Taken biological samples on patients with Autism Spectre Disorders
  Interventions: Other: Samples
- Healthy volunteers: Taken biological samples on patients healthy volunteers
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — Urinary and faecal samples

SUMMARY:
Autism Spectrum Disorder refers to complex neuro-developmental disorders that affect social communication and behavioral adaptation. Currently, the diagnosis of Autism Spectrum Disorder is based on a clinical examination that is performed classically during the first three years of life. The heterogeneity of the disorders occurring in autism make pathologies difficult to diagnose and manage.

The overall goal of this project is the identification of metabolic biomarkers based on clinical profile. The best characterization of physiopathological pathways will ultimately allow the identification of subgroups of subjects and facilitate the development of targeted therapeutics.

The proposed work aims to test the hypothesis of a disruption of tryptophan metabolism in Autism Spectrum Disorder via the gut microbiota.

DETAILED DESCRIPTION:
Autism Spectrum Disorder refers to complex neuro-developmental disorders that affect social communication and behavioral adaptation. In France, Autism Spectrum Disorderaffects about 1 in 100 people according to international criteria and is diagnosed in early childhood. Currently, the diagnosis of Autism Spectrum Disorder is based on a clinical examination that is performed classically during the first three years of life. The heterogeneity of the disorders occurring in autism make pathologies difficult to diagnose and manage.

The overall goal of this project is the identification of metabolic biomarkers based on clinical profile (based on behavioral and cognitive markers). The best characterization of physiopathological pathways (from the molecular scale to the phenotypic scale) will ultimately allow the identification of subgroups of subjects and facilitate the development of targeted therapeutics.

The proposed work aims to test the hypothesis of a disruption of tryptophan metabolism in Autism Spectrum Disorder via the gut microbiota.

ELIGIBILITY:
Inclusion Criteria (patient):

* 3-12 year old child
* Diagnosis of Autism Spectrum Disorders according to the DSM-5 (2013), invasive developmental disorder according to the ICD-10 (1993) or Autism Spectrum Disorders according to ICD-11 (2018)
* Affiliate or beneficiary of a social security scheme
* Consent signed by at least one of the parents

Exclusion Criteria (patient):

* Chronic inflammatory pathology
* Probiotic intake
* Taking medication (except melatonin) within 6 days before inclusion and until biological samples are collected

Inclusion Criteria (healthy volunteer):

* 3-12 year old child
* Affiliate or beneficiary of a social security scheme
* Consent signed by both parents

Exclusion Criteria (healthy volunteer):

* Chronic inflammatory pathology
* Digestive pathology
* Probiotic intake
* Taking medication within 6 days before inclusion and until biological samples are collected
* Personal and / or family history of neurological disease, epilepsy, psychiatric disorder, neurodevelopmental disorder, language disorder, overdrive, intellectual disability

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 3-12 year old children with and without Autism Spectrum Disorders
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
Urinary concentrations of tryptophan metabolites | At baseline
  Quantification by High-Performance Liquid Chromatography and Mass Spectrometry
Faecal concentrations of tryptophan metabolites | At baseline
  Quantification by using High-Performance Liquid Chromatography and Mass Spectrometry

SECONDARY OUTCOMES:
Characterization of gut microbiota | At baseline
  Characterization by 16S ribosomal RNA sequencing
Correlation of metabolic profiles of tryptophan and microbiotic profiles | At baseline
  Study of correlations from the outcomes measures 1, 2 and 3

CONTACTS AND LOCATIONS:
Overall Officials: Patrick EMOND, MD, Study Director — University Hospital, Tours
Locations (2):
- France (2):
  - Child psychiatry department, University Hospital, Tours, Tours
  - Clinical investigation center, University Hospital, Tours, Tours